CLINICAL TRIAL: NCT03975972
Title: Differences in Reading Achievement When Using Occupational-therapy Based Strategies Versus Standard Classroom-based Reading Intervention for Elementary School Children-a Pilot Study.
Brief Title: Occupational Therapy-based Literacy Intervention and Classroom Based Literacy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Turquessa Francis, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study00003591
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational Therapy Based Literacy Intervention (Experimental): For the intervention group, the results from the Inventory of Reading Occupations will be utilized to determine a prescriptive weekly intervention for each participant in the intervention group that will be provided to teachers based on student interest and literacy need. For the intervention group, each participant will be provided with a list of 12 questions that will be used to inform the intervention plan based on the interests of each participant within the intervention group. Collectively, the information from the 12 questions and the results of the Inventory of Reading Occupations will be used to determine a 9-week intervention plan for each participant within the intervention group. The researchers will work with the subjects twice per week, 30 minutes per session in the classroom using the prescriptive intervention that was determined from the assessments utilized.
  Interventions: Other: Occupational Therapy Based Literacy Intervention
- Standard Classroom Based Literacy Intervention (No Intervention): The control group will receive the standard reading instruction provided within the school. With the control group, the researchers will provide occupational therapy support to classroom teachers. But, will provide this support using the materials that are standardly provided within the classroom for literacy instruction. The researchers will provide support to the classroom teachers to students in the control group twice per week for 30 mintues per session in the classroom.

INTERVENTIONS:
Other: Occupational Therapy Based Literacy Intervention — Use of an occupational therapy-based literacy intervention that utilizes student interest to guide a prescriptive literacy intervention. Addressing reading as an occupation and making the necessary modifications to the literacy task to allows for increased engagement in the task. Increased engagement in literacy tasks, allows for opportunities to work on literacy deficit areas to address proficiency with reading ability.
  Arms: Occupational Therapy Based Literacy Intervention

SUMMARY:
The purpose of this study is to determine the impact of a literacy focused occupational therapy intervention program versus standard classroom-based reading intervention on reading engagement and reading achievement in elementary school-aged children with emotional disturbances.

DETAILED DESCRIPTION:
The elementary school will assist with recruitment by sending recruitment packets home to parents/legal guardian of children to consent to participation in the study. Interested families will return the signed consent form to the researchers in a sealed envelope. These signed consent forms will be collected from the school by the researchers. For children where a consent was provided by a parent or legal guardian, an assent form will be completed by the child for the child to also consent to participating the study, a requirement to ensure that the child has a choice in partaking in the study.

Once all consents have been received, all consenting student participants will be placed in either a control group or intervention group based on the students' classroom teacher. Both the control group and intervention group will be assessed using the Inventory of Reading Occupations(IRO) to determine their access to reading materials and their perceived proficiency with the reading tasks. Both the control group and intervention group's reading level will be obtained from the classroom teacher using the results of the Independent Reading Level Assessment® Framework (IRLA) from the beginning of the school year.

The intervention group will be provided with a 12-question survey to determine reading interest to guide the 9-week literacy intervention plan and ensure that the literacy intervention plan is in line with the IRLA reading Program. The control group will receive literacy instruction as proposed by the IRLA reading program and will not receive a specific occupation-based literacy intervention plan. Both the control and intervention group will have the principal investigator and student researchers available to provide one-on-one support during literacy instruction, with the intervention group receiving a specific literacy intervention plan while the control group continues with the literacy instructional material provided within the IRLA assessment framework. At the end of 9-weeks, the control group and intervention group will be re-administered the Inventory of Reading Occupations(IRO) and an updated reading achievement will be obtained from teacher from the student's scores on the Independent Reading Level Assessment® Framework (IRLA) at the end of the 9-week intervention period. The control group and intervention group's IRO and IRLA scores will be analyzed to find out the differences between the groups in reading interest, perceived reading proficiency and reading achievement. The researchers will be available by phone or email throughout the entirety of the study should questions arise about the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in grades 1-5 .
* Participants must be between the ages of 5-13 years of age: (the age is capped at a higher level due to the population this school serves where students may repeat a grade. So, the student may be older than most elementary aged children, but from a literacy perspective, they are functioning below their peers).
* Participants must be at least one grade level below peers in reading using assessment that is utilized in school.
* Participants must be able to speak English

Exclusion Criteria:

* Students who are unable to speak or read English due to assessments being in English
* Students who fall outside of the age criterion listed above
* Students that are on grade level with reading

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Reading Achievement | 9 weeks
  The reading level of student using the reading assessment that is utilized by the school: Independent Reading Level Assessment Framework (IRLA)

SECONDARY OUTCOMES:
Literacy Engagement | 9 weeks
  The amount of methods that the students using to access text, literacy tasks that the student engages in and the student's perceived proficiency with methods of accessing text. The Inventory of Reading Occupations (IRO) will be used to determine these three areas.

CONTACTS AND LOCATIONS:
Overall Officials: Turquessa Francis, Ed.D, Principal Investigator — SUNY Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be made available to other researchers.

REFERENCES:
- [Background] Grajo, L.C. & Candler, C. (2014). Children with reading difficulties: how occupational therapy can help. OT Practice, 19(13), 16-17.
- [Background] Grajo, L.C. & Candler, C. (2016). An occupation and participation approach to reading intervention (OPARI) part I: defining reading as an occupation. Journal of Occupational Therapy, Schools, & Early Intervention, 9(1), 74-85.
- [Background] Grajo LC, Candler C, Bowyer P, Schultz S, Thomson J, Fong K. Determining the Internal Validity of the Inventory of Reading Occupations: An Assessment Tool of Children's Reading Participation. Am J Occup Ther. 2016 May-Jun;70(3):7003220010p1-9. doi: 10.5014/ajot.2016.017582. PMID 27089292
- See also: American Occupational Therapy Association. The role of occupational therapy with literacy. — https://www.aota.org/Practice/Children-Youth/literacy.aspx